CLINICAL TRIAL: NCT02897843
Title: The Effect of Transcranial Direct Current Stimulation on Cognitive Side Effects of Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Raphael Braga, Psychiatrist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS16-0241
Record Dates: First submitted 2016-08-02; First posted 2016-09-13 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Depressive Disorder
Keywords: Electroconvulsive Therapy; Transcranial Direct Current Stimulation; cognition
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS (Sham Comparator): Sham tDCS sessions will last 20 minutes, but a real stimulus of 2 milliamps (mA) will be applied only during the first minute
  Interventions: Device: sham tDCS
- tDCS (Experimental): 20 minute tDCS sessions
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — tDCS stimulation will involve ten 20 minute stimulations daily, characterized by 2 milliamps (mA) anode over the left dorsolateral prefrontal cortex (DLPFC), with the cathode placed over the right suborbital region.
  Arms: tDCS
Device: sham tDCS — sham tDCS
  Arms: sham tDCS

SUMMARY:
Electroconvulsive therapy (ECT) is an effective treatment for a variety of psychiatric disorders. However, despite continued advances in ECT technique, neurocognitive dysfunction continues to be a frequent adverse effect. Declarative memory and less so selective memory are often impaired after an ECT course. Immediate memory, however, is broadly preserved. It is hypothesized that memory impairments are due to ECT induced disruptions on long term potentiation as well as in cerebral flux and glutamatergic and cholinergic systems. Different pharmacological agents for the treatment of ECT induced cognitive dysfunction have been tried. Agents such as opioids, vasopressin, neuropeptides, cholinergic agents, thyroid hormone, and stimulants have been used with equivocal results, and no controlled studies showed clear efficacy.

Transcranial direct current stimulation (tDCS) is a non-invasive, painless brain stimulation treatment that uses direct electrical currents to stimulate specific parts of the brain. Electrical currents are applied constantly at low intensities (1-2 mA) over a long period, usually in minutes (5-30 minutes), to achieve changes in cortical excitability by influencing spontaneous neural activity. There are two types of stimulation with tDCS: anodal and cathodal stimulation. Anodal stimulation acts to excite neuronal activity while cathodal stimulation inhibits or reduces neuronal activity. Several studies demonstrated moderate to strong effect sizes of tDCS in various neurocognitive and neuropsychiatric settings. Majority of studies show positive effects of tDCS on cognitive functioning among healthy volunteers and subjects with neurological or psychiatric conditions. Beneficial effects of online stimulation applied over the left dorsolateral prefrontal cortex have been reported for working memory, attention and information processing in depressed patients. To the investigators' knowledge no studies have evaluated the potential efficacy of tDCS for the prevention of ECT induced cognitive adverse effects.

In the current study, the investigators propose a double blind, randomized controlled trial to test the use of tDCS as a strategy to prevent or mitigate the memory impairments frequently associated with an ECT course.

DETAILED DESCRIPTION:
This is a prospective, random assignment, double blind, parallel group study with an adaptive design comparing the efficacy of tDCS performed during the course of ECT to that of sham tDCS in patients with a major depressive episode being treated with ECT. The investigators intend to recruit patients who are scheduled to receive an acute course of ECT. Patients who are able and willing to provide written informed consent, and who meet study criteria when screened, will be randomly assigned on a 1:1 ratio to receive a course of real tDCS or sham tDCS. Subjects will receive a standard acute course of bifrontal ECT (3X/week) and depressive symptomatology will be monitored with the Hamilton Rating Scale for Depression (HRSD-24) before each treatment.

The primary outcome will be change in cognition from baseline to end of study. The investigators will monitor cognitive changes before and after each ECT treatment, at the end of the treatment course and two months after the last treatment.

Secondary outcome will be the number of treatments needed to achieve remission. Remission is defined as two consecutive Hamilton Rating Scale for Depression (HRSD) scores <= 10, and HRSD total score does not change > 3 points or remains < 6 at the last two consecutive treatments. In addition, the investigators will collect data on other treatment parameters such as seizure duration, electroencephalogram (EEG) morphology as well as hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and above;
* Diagnosis of Major Depression confirmed by Structured Clinical Interview for Diagnostic and Statistical Manual IV (SCID-IV) interview;
* ECT is clinically indicated;
* Patient is competent to provide informed consent;

Exclusion Criteria:

* Lifetime DSM-IV diagnosis of schizophrenia, schizoaffective disorder or any other primary psychotic disorder as well as Bipolar Disorder, as defined in the DSM-IV;
* Current diagnosis of delirium or any major or minor neurocognitive disorder;
* Diagnosis of Mental Retardation;
* Limited English proficiency;
* Baseline Mini Mental State Exam (MMSE) score < 21 or a total score falling two standard deviations below the age- and education-adjusted mean, whichever is less;
* Skin lesions at the site of electrodes and any documented head or neck dermatological disorder;
* Person with any kind of neurostimulator, an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system;
* Any active general medical condition or central nervous system (CNS) disease which can affect cognition or response to treatment;
* A history of medication-resistant epilepsy in the family, and/or past history of seizures or unexplained spells of loss of consciousness during the previous 36 months
* Current (within the past three months) diagnosis of active substance dependence, or active substance abuse within the past week, as determined by interview and chart review.
* Active suicidal ideation, as measured by scores of 3 or more on item 3 of the HRSD;
* ECT within six months;
* The presence of any known or suspected contraindication to methohexital including but not limited to known allergic reactions to these agents, uncontrolled hypertension, arrhythmia, severe coronary artery disease and porphyria;
* Pregnancy as determined by interview and blood work done for ECT workup;
* Women who are breastfeed as determined by self-report;
* Status 4 or greater according to the criteria of the American Society of Anesthesiologists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Change in memory function | up to three months
  Change in memory function will be determined by a factor analysis of all memory tests

SECONDARY OUTCOMES:
Number of ECT treatments needed to achieve remission | up to three weeks
  Remission is defined as two consecutive Hamilton Rating Scale for Depression (HRSD) scores <= 10, and HRSD total score does not change > 3 points or remains < 6 at the last two consecutive ECT treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Braga, MD, Principal Investigator — Northwell Health
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided